CLINICAL TRIAL: NCT04808089
Title: The Feasibility of Asthma Application of Mobile Phone and Mobile Spirometry for Home Monitor of Asthma Patients to Achieve Optimal Asthma Control
Brief Title: The Feasibility of Asthma Application of Mobile Phone and Mobile Spirometry for Home Monitor of Asthma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ting-Yu Lin, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202100251B0
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Prospective randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Lung App. +ezOxygen (Experimental): Health Lung" App. (AstraZeneca Pharmaceuticals LP) is the application for mobile phone to help asthma care and is available freely in Google Play. Health Lung can be connected to the mobile spirometry, "ezOxygen" (Genius Holding Co.,Ltd Taiwan Branch).
  The functions of Health Lung App. include asthma control monitor, lung function monitor, controller and reliver inhaler reminder and recording, asthma educational topics in brief and information of air quality
  Subjects can get reminder to use inhaler on schedule, input ACT score to evaluate the asthma control, get education materials about asthma and operate spirometer to access lung function outside of hospital.
  he physicians in charge will get the information about control status score by ACT, adherence of controller and usage of reliver of patients between each clinical visit, if patients following the instruction of "Health Lung".
  Interventions: Other: Health Lung App. of mobile phone+ezOxygen mobile spirometry
- Usual care (Active Comparator): The research assistant assess/ teach inhaler technique, offering the asthma education as the regular clinical service.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Health Lung App. of mobile phone+ezOxygen mobile spirometry — Subjects can get reminder to use inhaler on schedule, input ACT score to evaluate the asthma control, get education materials about asthma and operate spirometer to access lung function outside of hospital.
  The physicians can get the information about control status, lung function, adherence of controller and usage of reliver of patients between each clinical visit, if patients following the instruction of "Health Lung".
  Arms: Health Lung App. +ezOxygen
Other: Usual care — The research assistant assess/ teach inhaler technique, offering advice on adherence, delivering patient self-management asthma action plan and education the meaning of asthma control accessed by ACT.
  Arms: Usual care

SUMMARY:
The aim of the present study is to explore if the "Health Lung" application of smart phone and portable spirometry "ezOxygen" can further improve asthma control for chronic asthma adult patients with well asthma control (ACT 20~24, but not 25), compared to hospital-based usual care in a medical center.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease. Despite we have academic treatment guidelines, and the asthma treatment develops persistently, many asthma patients do not have well control.

Asthma Control Test (ACT) is a patient self-administered tool for identifying those with poorly controlled asthma. ACT includes 5 items on 5-point scale, with 4-week recall on symptoms and daily functioning. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.

In addition to correct diagnosis and prescription by physicians, achieving asthma well control depend on the patient's ability of self- management.

The self-management of asthma patients includes monitor of symptoms, monitor of peak expiratory flow, compliance of inhaler and avoiding the asthma triggers.

Portable digital tools may be the possible solution for home monitor of asthma patients. Through the application of mobile phone and hand-held mobile spirometry, asthma patients can monitor their symptoms and lung function at home outside of hospital.(5-7)。

"Health Lung" (AstraZeneca Pharmaceuticals LP) is the application for mobile phone to help asthma care and is available freely in Google Play. Health Lung can be connected to the mobile spirometry, "ezOxygen" (Genius Holding Co.,Ltd Taiwan Branch).

Therefore, the functions of this App. include asthma control monitor, lung function monitor, controller and reliver inhaler reminder and recording, asthma educational topics in brief and information of air quality. The physicians can get the information about control status, lung function, adherence of controller and usage of reliver of patients between each clinical visit, if patients following the instruction of "Health Lung".

However, how the patients are willing to use digital tools at home and what is the real impact on the current hospital-based asthma care need to be validated.

The aim of the present study is to explore if the "Health Lung" application of smart phone and portable spirometry "ezOxygen" can further improve asthma control for chronic asthma adult patients with well asthma control (ACT 20~24, but not 25), compared to hospital-based usual care in a medical center.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 65 years old.
* Regular prescription of inhaled corticosteroid-containing medications at least 6 months.
* The asthma control is well but not in total control: ACT 20~24, but not to full score 25.

Exclusion Criteria:

* Patients were excluded if they do not have internet-connecting smart phone.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Asthma control | 3 months
  The improvement of asthma control evaluated by Asthma Control Test (ACT). The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.

SECONDARY OUTCOMES:
The compliance of controller | 3 months
  The adherence of asthma inhaler drugs will be evaluated by the questionnaire about inhaler compliance.
  According to your memory, how often did you forget to follow the doctor's order to use the inhaler(s) in the past 4 weeks?
  1.Almost every day; 2. No more than 7 days; 3. No more than 14 days; 4. More than 15 days
The satisfaction of digital tools in study group | 3 months
  The subjects in study arm will be asked about how they satisfy the functions of "Health lung" App. and ezOxygen spirometry via 100-mm length visual analogue scale. 0: the most dissatisfaction/unhelpful to 100 mm: the most satisfaction/helpful

OTHER OUTCOMES:
The impact of digital tools on clinical practice | 3 month
  The physicians in charge in study arm will be ask if they order any further exam or prescription due to the information provided by digital tools.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Lin, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan